CLINICAL TRIAL: NCT07115862
Title: Effect of Pomegranate Juice on Gut Inflammation, Quality of Life and the Gut Microbiome in Patients With Ulcerative Colitis: A Pilot Study
Brief Title: Effects of Pomegranate Juice on Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-25-1553; T32DK007180 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (Disorder)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will be consuming 237 ml of pomegranate juice for the first 8 weeks of the study and their habitual diet without pomegranate juice for the second 8 weeks
  Interventions: Other: pomegranate juice -> habitual diet
- Delayed start (Experimental): Participants in this arm will consume their habitual diet for the first 8 weeks of the study and drink 237 ml of pomegranate juice for the second 8 weeks
  Interventions: Other: habitual diet -> pomegranate juice

INTERVENTIONS:
Other: pomegranate juice -> habitual diet — 237 ml of pomegranate juice for the first 8 weeks -> habitual diet for the second 8 weeks
  Arms: Intervention
Other: habitual diet -> pomegranate juice — habitual diet for the first 8 weeks -> 237 ml of pomegranate juice for the second 8 weeks
  Arms: Delayed start

SUMMARY:
The purpose of this study is to determine whether consumption of 237 ml of pomegranate juice daily for 8 weeks will:

1. lower inflammation (in the gut as well as generally in the body) and improve your overall quality of life
2. affect the microbes living in the gut (gut microbiota)

DETAILED DESCRIPTION:
the study is aimed at evaluating the effects of pomegranate juice (PomJ) on: 1) gut inflammation (fecal calprotectin and Simple Clinical Colitis Activity Index) and quality of life; 2) circulating inflammatory markers (e.g., hs-CRP, IL-6, IL-10, TNF-a, IL-1b, IL-8, LBP, LPS) and markers of oxidative stress (blood and urine malondialdehyde (MDA)) and 3) gut microbiota composition and functionality (urinary and circulating urolithin metabolites, fecal SCFAs/BAs, blood LBP and LPS, etc.). We will perform a randomized, controlled, 16-week trial to generate preliminary evidence on the effects of PomJ consumption in patients with mild-to-moderate UC. Participants will be randomly assigned to one of two groups: intervention group and delayed start group. The study will involve 2 phases, each lasting for 8 weeks. During Phase 1, the intervention group will consume 237 ml of PomJ daily, while the delayed start group will follow their habitual diet. Data generated from the delayed start group during Phase 1 will serve as the control for the study. During Phase 2, the intervention group will stop consuming PomJ and switch to consuming their habitual diet, while the delayed start group will consume 237 ml of PomJ daily for 8 weeks. Data generated from the intervention group during Phase 2 will serve as a follow-up to explore whether the effects of PomJ consumption persist after consumption is stopped (this will be an exploratory outcome).

ELIGIBILITY:
Inclusion Criteria:

* • Adults ≥ 18 yo

  * Following a low-polyphenol and fiber diet (< 3 servings of fruits/vegetables per day)
  * Mild-to-moderate UC at the time of screening (2 ≤ partial Mayo scores ≤ 5)
  * Supportive evidence of active inflammation (hsCRP >1 mg/L, fecal calprotectin >50 µg/g stool, or abnormal lower endoscopy) in individuals with biopsy-proven UC
  * Patients on 5-aminosalicylates must be on a stable dose for ≥ 4 weeks prior to screening
  * Patients on treatment with immunosuppressive therapy (e.g., azathioprine/6-mercaptopurine, methotrexate) must be on stable dose for 8 weeks prior to baseline visit
  * At the time of baseline visit, patients may be on no more than 20 mg/day of prednisone and 9 mg/day of budesonide MMX
  * Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* • Non-English speaker

  * Vegetarian/vegan
  * Known pomegranate allergy
  * Documented chronic disease besides UC, including diabetes, renal or liver diseases, metabolic syndrome, active cancer, MI or stroke, history of gastric bypass
  * Patients with CD, indeterminate/severe to fulminant colitis
  * History of colectomy or colonic dysplasia
  * Presence of ileal pouch or ostomy
  * Evidence of active bacterial or viral gastroenteritis as indicated by positive stool studies for ova & parasites, Clostridium difficile, and stool culture
  * Recent hospitalizations (within 2 weeks of screening) for UC requiring IV steroids
  * Presence of the following labs indicative of severe colitis: a. Hemoglobin < 8.0 g/dl b. Albumin < 3.0 g/dl
  * Recent systemic antibiotics use (within 3 months of screening) or active use of anti-diarrheal medications
  * Taking supplements known to affect metabolism or gut microbiota composition (probiotics, fiber, etc.), unless willing to stop for the study duration
  * Use of Total Parenteral Nutrition (TPN)
  * Use of cyclosporine, tacrolimus, or thalidomide within 2 months prior to screening
  * Taking exogenous hormones (e.g., hormone replacement therapy)
  * Recent weight fluctuations (>10% in the last 6 months)
  * Smoker or living with a smoker
  * Use of >20 g of alcohol per day
  * Unable or unwilling to comply with the study protocol (including unwillingness to avoid watermelon and other lycopene-rich foods for the whole duration of the study)
  * Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
simple clinical colitis activity index (SCCAI) | At baseline, 8 weeks and 16 weeks
  Simple Clinical Colitis Activity Index (SCCAI) includes questions about bowel frequency, urgency of defecation, etc. Measured by the number of points/scores.
Fecal calprotectin | At baseline, 8 weeks and 16 weeks
  To evaluate effects of PomJ on gut inflammation in patients with mild-to-moderate UC. The primary outcome will be levels of fecal calprotectin (objective measure). Fecal calprotectin levels will be assessed via a commercially available ELISA kit in mcg/g.

SECONDARY OUTCOMES:
Biomarkers of inflammation and oxidative stress | At baseline, week 8 and week 16
  Blood interleukin-6 (IL-6) in pg/ml
Biomarkers of inflammation and oxidative stress | At baseline, week 8 and week 16
  Blood interleukin-10 (IL-10) in pg/ml
Biomarkers of aging and oxidative stress | At baseline, week 8 and week 16
  Blood TNF-a in pg/ml
Biomarkers of inflammation and oxidative stress | At baseline, week 8 and 16
  Blood IL-1b in pg/ml
Biomarkers of inflammation and oxidative stress | At baseline, weeks 8 and 16
  Blood IL-8 in pg/ml
Biomarkers of inflammation and oxidative stress | At Baseline, weeks 8 and 16
  Blood hs-CRP in mg/ml
Biomarkers of inflammation and oxidative stress | At baseline, weeks 8 and 16
  Urine malondialdehyde (MDA) in ng/ml
Biomarkers of inflammation and oxidative stress | At baseline, weeks 8 and 16
  Blood MDA in nmol/ml
Biomarkers of inflammation and oxidative stress | At baseline, weeks 8 and 16
  Urine 8OHdG in ng/mg
Biomarkers of inflammation and oxidative stress | At baseline, weeks 8 and 16
  Blood 8OHdG in ng/ml

OTHER OUTCOMES:
Gut-derived metabolites | At baseline, weeks 8 and 16
  Blood urolithin metabolites in micromoles/L
Gut-derived metabolites | At baseline, weeks 8 and 16
  Urine urolithin metabolites
Microbial inflammatory components | At baseline, weeks 8 and 16
  Blood lipopolysaccharide in ng/ml
Microbial inflammatory components | At baseline, weeks 8 and 16
  Blood LPS binding protein in micrograms/ml
Microbial-derived metabolites | At baseline, weeks 8 and 16
  Fecal short-chain fatty acids (SCFAs) in micromoles/g
Microbial-derived metabolites | At baseline, weeks 8 and 16
  Fecal bile acids (BAs) in ng/ml
Gut microbiota composition | At baseline, weeks 8 and 16
  The stool specimen will be collected by the participants at home at baseline and week 12 utilizing our Stool Collection Kit as per instructions. Immediately after collection, the specimen will be frozen in a home freezer and delivered in an insulated container to the UCLA Center for Human Nutrition. At UCLA, the specimen will be stored at - 80 ºC. Fecal microbiological analyses. Approximately 1g of the stool will be weighed and dried in a vacuum drying oven (15 in Hg) at 80 ºC for 48 hours, then weighed again to establish the moisture content so that all counts can be corrected to dry weight. From another aliquot of remaining fecal samples, DNA will be extracted using bead beating with a commercial extraction system (DNeasy PowerSoil® DNA Isolation Kit, Qiagen, Valencia, CA). The quality of the DNA samples will be confirmed using a Nanodrop 1000 (Thermo Fisher Scientific, Wilmington, DE). Extracted DNA will be transferred to UCLA Microbiome Core facility for MiSeq sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - West Los Angeles VA Medical Center, Los Angeles, California
  - UCLA Center for Human Nutrition, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
Data analysis will be performed in-house.